CLINICAL TRIAL: NCT01890889
Title: A Double-blinded, Placebo-controlled Randomized Trial Assessing the Extent to Which Consumption of Two Different Amounts of a Non-Pharmaceutical Food Supplement Can Improve Cardiovascular Health
Brief Title: Study of Changes in Total Cholesterol Levels as a Function of Consuming a Supplement Designed to Improve Cardiovascular Health
Acronym: AdBiotech
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Health Technologies, Inc. (Network)
Responsible Party: Principal Investigator, Gilbert R Kaats, Dr. Gilbert R. Kaats, PhD, Integrative Health Technologies, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 065
Record Dates: First submitted 2013-06-27; First posted 2013-07-02 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Cholesterol; Hyperlipidemia; Hypercholesteremia
Keywords: Total Cholesterol; LDL
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ad-Chol-Pre (Active Comparator): A functional food ingredient designed to inhibit cholesterol absorption. ACP is a freeze dried defatted egg powder containing specific Anti-NPCIL1 (Niemann-Pick C1-like 1) IgY. NPC1L1 is known as a biological target of the cholesterol-uptake inhibitor, Ezetimibe.
  Interventions: Dietary Supplement: Ad-Chol-Pre
- Half-dose Ad-Chol-Pre (Active Comparator): A half-dose of the active comparator in arm one is administered. A functional food ingredient designed to inhibit cholesterol absorption. ACP is a freeze dried defatted egg powder containing specific Anti-NPCIL1 (Niemann-Pick C1-like 1) IgY. NPC1L1 is known as a biological target of the cholesterol-uptake inhibitor, Ezetimibe.
  Interventions: Dietary Supplement: Half-dose Ad-Chol-Pre
- Capsule containing inactive component of defatted egg yolk (Placebo Comparator): Placebo capsule is filled with defat egg yolk only without specific IgY which is anti-NPC1L1 IgY, designed to look and taste the same as the active product capsule, but does not contain the active component.
  Interventions: Other: Defatted egg yolk without the active ingredient of the other two interventions

INTERVENTIONS:
Dietary Supplement: Ad-Chol-Pre
  Other Names: Anti-NPC1L1 IgY; Ezetimibe
  Arms: Ad-Chol-Pre
Dietary Supplement: Half-dose Ad-Chol-Pre
  Other Names: Ad-Chol-Pre; Anti-NPC1L1 IgY; Ezetimibe
  Arms: Half-dose Ad-Chol-Pre
Other: Defatted egg yolk without the active ingredient of the other two interventions
  Other Names: Capsule manufactured to mimic the Ad-Chol-Pre capsule, only not containing the active component.
  Arms: Capsule containing inactive component of defatted egg yolk

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a food-source nutrient containing bitter orange by comparing changes 45 blood chemistries and self-reported quality of life.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of a food-source nutrient by comparing changes in total cholesterol levels, 44 other blood chemistries, and self-reported quality of life as a function of consuming two different functional-food supplements versus a placebo in a 60-day study.

Upon completion of the pre-study screening, and after having received an explanation of the requirements, risks and benefits, and completing the informed consent interview with the research coordinator, subjects will execute a written informed consent. Subjects will be randomly assigned to one of three study groups.

Relevant Background Information.

A factor leading to development of vascular disease, a leading cause of death in industrialized nations, is elevated serum cholesterol. It is estimated that 19% of Americans between the ages of 20 and 74 years of age have high serum cholesterol. However, in an analysis of 10,000 test results in our database from subjects similar to those who are likely to participate in this study, we found 37% of subjects had TC scores between 200 and 250 and 10.3% above 250.

The most prevalent form of vascular disease is arteriosclerosis, a condition associated with the thickening and hardening of the arterial wall. The regulation of whole-body cholesterol homeostasis involves the regulation of intestinal cholesterol absorption, cellular cholesterol trafficking, a modulation of cholesterol biosynthesis, bile acid biosynthesis, steroid biosynthesis and the catabolism of the cholesterol-containing plasma lipoproteins. Regulation of intestinal cholesterol absorption has proven to be an effective means by which to regulate serum cholesterol levels.

Ad-Chol-Pre (ACP) is a functional food ingredient designed to inhibit cholesterol absorption. ACP is a freeze dried defatted egg powder containing specific Anti-NPCIL1 (Niemann-Pick C1-like 1) IgY. NPC1L1 is known as a biological target of the cholesterol-uptake inhibitor, Ezetimibe. In previous unpublished pilot studies examining the safety and efficacy of ACP include:

* ACP was shown to produce a statistically inhibition of [3H]-Cholesterol absorption from 50 ug/ml (P<0.05) in NPC1L1 over-expressing HepG2 cell lines as compared to an inhibition of 10ug/ml with Ezetimibe alone.
* I preliminary unpublished animal studies, ACP was shown to significantly inhibit radiolabelled cholesterol. ACP was found to significantly lower total cholesterol (38% ~56%) and LDL cholesterol (46~57%) in bloods from animals fed who had been fed a high fat diet for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* be an English-speaking male or female at least 18 years of age;
* have a total cholesterol level between 200 mg/dL and 250mg/dL
* have a LDL level between 100 mg/dL and 160 mg/dL
* not have allergic reactions to eggs or egg products
* not have consumed cholesterol-lowering drugs within 2 months of starting the study
* agree to follow the requirements of the study as set forth in this Informed Consent
* agree to withdraw from the study if becoming pregnant during the study.

Exclusion Criteria:

* do not speak English;
* are under 18 years of age;
* have a total cholesterol level below 200 mg/dL or above 250 mg/dL
* have a LDL level below 100 mg/dL or above 160 mg/dL
* have allergic reactions to eggs or egg products
* have consumed cholesterol-lowering drugs within 2 months of starting the study
* are pregnant or nursing;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Total Cholesterol and LDL levels at 30 days | 0 and 30 days
Change from baseline in Total Cholesterol and LDL levels at 60 days | 0 and 60 days
Change from mid-point in Total Cholesterol and LDL levels at 60 days | 30 and 60 days

SECONDARY OUTCOMES:
Blood Chemistry Measurements | 0, 30, and 60 days
  Remaining lipids, Complete Blood Count, Metabolic Panel, Thyroid Stimulating Hormone, Cardio C-reactive Protein
Self-reported Quality of Life | 0, 30, and 60 days
Number of participants with adverse effects | up to 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert R Kaats, PhD FACN, Principal Investigator — Integrative Health Technologies, Inc.; Harry G Preuss, MD MACN, Study Chair — Georgetown University Medical Center, Dept of Biochemistry, Medicine and Pathology; Sidney J Stohs, PhD, Study Director — Dean Emeritus, Creighton University Health Sciences Center
Locations (1):
- Integrative Health Technologies, San Antonio, Texas, United States